CLINICAL TRIAL: NCT00110513
Title: A Multicenter, Multinational Study to Assess the Safety and Efficacy of Antithrombin Alfa in Hereditary Antithrombin (AT) Deficient Patients in High-Risk Situations for Thrombosis
Brief Title: Recombinant Human Antithrombin (rhAT) in Patients With Hereditary Antithrombin Deficiency Undergoing Surgery or Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: rEVO Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GTC AT HD 012-04
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Antithrombin III Deficiency
Keywords: Antithrombin Deficiency, Congenital or Hereditary; Antithrombin III Deficiency; ATIII; Hereditary Antithrombin Deficiency (HD)
MeSH Terms: conditions — Antithrombin III Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant Human Antithrombin (rhAT) Infusion (Experimental): Intravenous infusion of rhAT.
  Interventions: Biological: Recombinant human antithrombin (rhAT)

INTERVENTIONS:
Biological: Recombinant human antithrombin (rhAT) — Up to 24 hours prior to the scheduled elective surgical procedure, caesarean section, or delivery induction, each patient will receive an initial intravenous loading dose followed by a continuous intravenous infusion of recombinant human antithrombin (rhAT) that will target and maintain an AT activity that is > 80% and < 120% of normal. The dosing objective for all study patients is maintenance of the AT activity at > 80% and < 120% of normal during the high-risk period for thromboembolic events. Dosing and dose adjustments will be based on the results of AT activity determinations performed prior to and during treatment.
  Other Names: Recombinant human antithrombin (Tradename: ATryn)

SUMMARY:
Patients with hereditary antithrombin deficiency are at increased risk of venous thrombosis and pulmonary embolism, particularly during certain high risk procedures. The trial focused on patients with confirmed hereditary antithrombin deficiency who were undergoing a surgical procedure or induced/spontaneous labor and delivery, and/or caesarean section. The study assessed the incidence of thromboembolic events following prophylactic intravenous administration of recombinant human antithrombin (rhAT) to patients with hereditary antithrombin (AT) deficiency in situations usually associated with a high risk for thromboembolic events.

DETAILED DESCRIPTION:
GTC Biotherapeutics established clinical trial sites in Europe, Canada, Australia, Austria and Canada. GTC Biotherapeutics provided an international clinical team to support site registration requirements once a patient was identified for treatment. GTC Biotherapeutics also provided consultation to help evaluate patient eligibility.

In September 2006, GTC Biotherapeutics modified exclusion criteria 1 (below) to allow for the participation of previously excluded patients with the hereditary thrombophilic disorders Factor V Leiden and prothrombin gene mutation (G20210A).

ELIGIBILITY:
Inclusion Criteria:

1. Have hereditary antithrombin deficiency (HD) with a personal history of venous thromboembolic events.
2. Have a history of HD that includes 2 or more plasma AT activity values ≤ 60%.
3. Be scheduled to have an elective procedure(s) known to be associated with a high risk for occurrence for DVT. This will include non-pregnant surgical patients or pregnant patients scheduled for caesarean section or delivery induction.
4. Be at least 18 years of age, not exceeding 80 years of age.
5. Have signed an informed consent form.
6. Have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline. This applies only to female non-pregnant surgical patients of childbearing potential.
7. Are able to comply with the requirements of the study protocol.

In addition, hospitalized pregnant HD patients in active labor and eligible HD patients previously treated with rhAT were allowed entry into the study.

Exclusion Criteria:

1. Patients who have a diagnosis of another hereditary thrombophilic disorder (e.g. activated protein C(APC) resistance/Factor V Leiden, Protein S or C deficiency, prothrombin gene mutation (G20210A), or acquired (lupus anticoagulant) thrombophilic disorder).
2. Patients who have a baseline bilateral ultrasound positive for acute DVT or baseline diagnostic testing (if required) that is positive for a thromboembolic event other than acute DVT.
3. Patients who have a known allergy to goats or goat products.
4. Patients who have participated in a study employing a different investigational drug within 30 days of the start of their participation in the current trial.
5. Patients using fondaparinux sodium or the oral thrombin inhibitor, ximelagatran, or are expected to be treated with fondaparinux sodium or ximelagatran during the study period (up to 7 days after stop of treatment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Tait, MD, Principal Investigator — Glasgow Royal Infirmary
Locations (17):
- United States (3):
  - New Haven, Connecticut
  - St Louis, Missouri
  - New York, New York
- North Gosford, Australia
- Vienna, Austria
- Canada (2):
  - Ottawa, Ontario
  - Vancouver
- Montpellier, France
- Berlin, Germany
- Alessandria, Italy
- United Kingdom (7):
  - Exeter, Devon
  - Chichester, West Sussex
  - Cambridge
  - Glasgow
  - London
  - Nottingham
  - Plymouth

REFERENCES:
- [Derived] DeJongh J, Frieling J, Lowry S, Drenth HJ. Pharmacokinetics of recombinant human antithrombin in delivery and surgery patients with hereditary antithrombin deficiency. Clin Appl Thromb Hemost. 2014 May;20(4):355-64. doi: 10.1177/1076029613516188. Epub 2013 Dec 11. PMID 24335249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included non pregnant patients who were scheduled for surgery and pregnant patients who were scheduled for caesarean section or delivery induction or were hospitalized in active labor.
Pre-assignment Details: Eighteen patients were treated with recombinant human antithrombin (rhAT) and analyzed for safety.
Groups:
- Recombinant Human Antithrombin (rhAT) Infusion: Up to 24 hours prior to the scheduled elective surgical procedure, caesarean section, or delivery induction, each patient received an initial intravenous loading dose of recombinant human antithrombin (rhAT)followed by a continuous intravenous infusion dose of recombinant human antithrombin (rhAT) to maintain an antithrombin (AT) activity level of >80% and <120% of normal.
Period: Overall Study
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Region of Enrollment [Number; unit: participants]
  France | 3
  Canada | 2
  Australia | 1
  Germany | 1
  United Kingdom | 8
  Italy | 1
  United States | 2
Prior history of thromboembolism [Number; unit: Participants] | 18
Antithrombin (AT) activity level <60% [Number; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Thromboembolic Events Acute Deep Venous Thrombosis (DVT) and/or Thromboembolic Events Other Than Acute Deep Venous Thrombosis (DVT)
Description: To assess the incidence of thromboembolic events acute deep venous thrombosis (DVT) and/or thromboembolic events other than acute deep venous thrombosis (DVT) by clinical signs and symptoms of venous thromboembolism (VTE), confirmed by diagnostic assessments.
Time Frame: During treatment and follow up period of 7 days
Population: Intent to treat population
Measure: Number; unit: Participants
Groups:
- Recombinant Human Antithrombin (rhAT) Infusion: Up to 24 hours prior to the scheduled elective surgical procedure, caesarean section, or delivery induction, each patient received an initial intravenous loading dose of recombinant human antithrombin (rhAT)followed by a continuous intravenous infusion dose of recombinant human antithrombin (rhAT) to maintain an antithrombin (AT) activity level >80% and <120% of normal.
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Number analyzed (Participants) | 18
Participants | 0

ADVERSE EVENTS:
Time Frame: Until 28 days after end of treatment.
Arm/Group | Recombinant Human Antithrombin (rhAT) Infusion
Serious Adverse Events (participants affected / at risk) | 5/18
Other Adverse Events (participants affected / at risk) | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Antithrombin (rhAT) Infusion (N=18)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Enterobacter Sepsis (Infections and infestations) | 1 (1)
Intra-Abdominal (Gastrointestinal disorders) | 1 (1)
DVT (Vascular disorders) | 1 (1) — An ultrasound of the lower extremities performed on post-operative day 14, revealed an occlusive thrombus in the right saphenous vein which was noted on previous ultrasound performed and had progressed to the popliteal vein. Reported as not related.
Hemoglobin decreased (Investigations) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — The patient received study drug from 21 November 2005 through 25 November 2005. On 09 December 2005, the patient experienced bilateral pulmonary embolism, which was reported as an important medical event and described as severe.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Antithrombin (rhAT) Infusion (N=18)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (5)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Oedema Peripheral (General disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Post Procedural Hemmorhage (Injury, poisoning and procedural complications) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Vaginal Laceration (Reproductive system and breast disorders) | 3 (3)
Haematoma (Vascular disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental Discomfort (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Feeling Hot (General disorders) | 1 (1)
Injection Site Bruising (Gastrointestinal disorders) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Incision Site Complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (1)
Wound Complicaton (Injury, poisoning and procedural complications) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1)
Hepatic Enzyme Abnormal (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Afterbirth Pain (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Nipple Pain (Reproductive system and breast disorders) | 1 (1)
Crackles Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphangitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No